CLINICAL TRIAL: NCT02641522
Title: Modulation of STAT3 Signaling With Siltuximab in Type 1 Diabetes
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Carla Greenbaum, MD (Other)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor-Investigator, Carla Greenbaum, MD, Director, Diabetes Program, Benaroya Research Institute
Organization: Benaroya Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EMU-002
Record Dates: First submitted 2015-12-23; First posted 2015-12-29 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Type 1 Diabetes
Keywords: T1D; Type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — siltuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Post-Infusion (Experimental): Single infusion of siltuximab (11 mg/kg)
  Interventions: Drug: Siltuximab

INTERVENTIONS:
Drug: Siltuximab — Single infusion of siltuximab (11 mg/kg)
  Other Names: Sylvant

SUMMARY:
The purpose of this study is to evaluate the effects of siltuximab on immune cell functions in patients with Type 1 diabetes (T1D).

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), single center, non-randomized (patients are not assigned by chance to treatment groups), Mechanistic Study (a study that focuses on the biologic activity of the drug, rather than on disease treatment). Up to 10 patients with Type 1 diabetes (T1D) will be enrolled in the study. Participants will receive a single dose of siltuximab and blood samples will be obtained a total of 6 times until 12 weeks after dosing. Cells will be isolated from the blood samples and used to measure specific activities of cells in the immune system. Safety evaluations for adverse events, clinical laboratory tests, vital signs, and physical examination will be performed throughout the study. The end of study is the date of the last assessment for the last patient.

ELIGIBILITY:
Inclusion Criteria:

1. Positive for at least one diabetes-related autoantibody any time since diagnosis, including by not limited to: Glutamate decarboxylase (GAD-65) Insulin, if obtained within 10 days of the onset of exogenous insulin therapy; IA-2; ZnT8
2. Peak stimulated C-peptide level ≥ 0.1 pmol/mL following a mixed meal tolerance test (MMTT) conducted within 60 days of enrollment
3. Females of child-bearing potential must be willing to use effective birth control and refrain from donating eggs for the purposes of assisted reproduction for duration of study.
4. A woman of childbearing potential must have a negative serum (β-human chorionic gonadotropin [β-hCG]) or urine pregnancy test at screening and prior to dosing.
5. During the study, and for 3 months after receiving the study agent, a woman must agree to not donate eggs (ova, oocytes) for the purposes of assisted reproduction.
6. Willing and able to give informed consent for participation.

Exclusion Criteria:

1. History of severe reaction or anaphylaxis to human, humanized or murine monoclonal antibodies;
2. History of malignancy or serious uncontrolled cardiovascular disease or hypertension, nervous system, pulmonary, renal, or gastrointestinal disease, or significant dyslipidemia despite therapy;
3. Any history of recent (within 3 months) serious bacterial, viral, fungal, or other opportunistic infections;
4. History or serologic evidence of current or past HIV, Hepatitis B, or Hepatitis C;
5. Positive QuantiFERON or PPD TB test, history of tuberculosis, or active TB infection;
6. Active infection with EBV ;
7. Active infection with CMV;
8. Diagnosis of liver disease or elevated hepatic enzymes, confirmed by repeat tests, as defined by ALT, AST, or both > 1.5 x the upper limit of age-determined normal (ULN) or total bilirubin > ULN;
9. Any of the following hematologic abnormalities, confirmed by repeat tests:

   * White blood count <3,000/μL or >14,000/μL
   * Lymphocyte count <500/μL
   * Platelet count <150,000 /μL
   * Hemoglobin <8.5 g/dL or > or = to 17 g/dL
   * Neutrophil count <2,000 cells/μL
10. Females who are pregnant or lactating;
11. Receipt of live vaccine (e.g. varicella, measles, mumps, rubella, cold-attenuated intranasal influenza vaccine, bacillus Calmette-Guérin, and small pox) in the 6 weeks before treatment;
12. Receipt of non-live vaccine in the 4 weeks before treatment;
13. Any medical or psychological condition that in the opinion of the Sponsor Investigator would interfere with the safe completion of the trial;
14. Receipt of an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 3 months or 5 half-lives before enrollment or is currently enrolled in the treatment stage of an investigational study;
15. Receipt of any immune-modulating biologic drug within 3 months of enrolling in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2017-03-16 (Actual); Study Completion 2017-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carla Greenbaum, MD, Principal Investigator — Benaroya Research Institute
Locations (1):
- Benaroya Research Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Siltuximab
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Siltuximab
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.1 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in IL-6 Stimulated Intracellular p-STAT3 at Week 12
Description: Change in IL-6 stimulated intracellular p-STAT3 between Week 12 and baseline
Time Frame: 0-to-12 weeks
Population: 1 participant was excluded from analysis because of technical problems with processing samples.
Measure: Mean (Standard Deviation); unit: Percent change from Baseline
Arm/Group | Siltuximab
Number analyzed (Participants) | 9
Percent change from Baseline | -4.31 (15.99)

2. Other Pre Specified Outcome: Adverse Event Monitoring
Description: Monitor adverse events associated with siltuximab treatment. All AE related to study drug will be tabulated along with their grade.
Time Frame: 0-to-12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 0-to-12 weeks
Arm/Group | Siltuximab
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Siltuximab (N=10)
Nuetrophil count decreased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Siltuximab (N=10)
Nuetrophil count decreased (Investigations) | 6
White blood cell decreased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 2
Hypoglycemia (Metabolism and nutrition disorders) | 1
Upper respiratory infection (Infections and infestations) | 3
Infections and infestations - Other - chalazion (Infections and infestations) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-23): https://cdn.clinicaltrials.gov/large-docs/22/NCT02641522/Prot_SAP_000.pdf